CLINICAL TRIAL: NCT00143767
Title: Magnetic Resonance Imaging of Brain Development in Attention Deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Other Study IDs: METC 05/036
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Magnetic Resonance Imaging
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The primary purpose of this study is to investigate brain whether ADHD represents a disruption or a delay of brain development. Children and adolescents both with and without ADHD are asked to participate in several MRI sessions, two years apart. This will allow us to chart brain development over time, both in typical development and ADHD, and therefore to address whether ADHD represents a disruption or a delay of typical brain development.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is a common and impairing neuropsychiatric disorder of childhood, occurring in 3 to 5% of all school-age children. This disorder is associated with greater risks for low academic achievement, school dropouts, poor family and peer relations, aggression, substance abuse, driving accidents and chronic problems in adult adaptation. As such, it has an enormous impact on the utilization of medical and health care services, and the direct and indirect costs of this disorder are high. However, in a large number of children symptoms dissipate as they grow up and they go on to function normally and lead typical lives. This has lead to speculation that ADHD may not so much represent a disruption, as a delay of brain development. This aim of this study is to address this issue.

There is a growing body of research supporting the existence of deficits in brain anatomy associated with ADHD, with evidence of reductions in overall brain size, cortical gray matter and subcortical structures. However, reported effect sizes are small and results not always consistent. Anatomical MRI studies may be easily confounded, as brain development is complex and associated with both progressive and regressive changes in brain anatomy. In this study, we propose to combine longitudinal data from a large cohort of children and adolescents with state-of-the-art imaging methods (including diffusion tensor imaging and voxelbased morphometry) to investigate brain development in ADHD. This will allow us to address the question whether ADHD represents a disruption or a delay of brain development.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 - 18 years at initial MRI

Inclusion Criteria for Subjects with ADHD:

* DSM-IV (APA, 1994) diagnosis of ADHD, according to DISC interview
* Scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form(TRF)

Inclusion Criteria for Controls:

* No DSM-IV (APA, 1994) diagnosis, according to DISC interview
* No scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)

Exclusion Criteria:

* IQ < 70
* Major illness of the cardiovascular, the endocrine, the pulmonal or the gastrointestinal system
* Presence of metal objects in or around the body (pacemaker, dental braces)
* History of or present neurological disorder
* For individuals over 12 years of age: legal incompetence, defined as the obvious inability to comprehend the information that is presented by the investigator and is outlined in the Information letter and on which the decision to participate in the study is to be based

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Durston, Ph.D., Principal Investigator — Rudolf Magnus Institute of Neuroscience, University Medical Center Utrecht; Herman van Engeland, M.D. Ph.D., Study Chair — Rudolf Magnus Institute of Neuroscience, University Medical Center Utrecht
Locations (1):
- Dept. of Child and Adolescent Psychiatry, UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: Lab homepage with info for subjects (in Dutch) — http://www.niche-lab.nl